CLINICAL TRIAL: NCT01902641
Title: Comparing Intubating Conditions and Patient Satisfaction Using Succinylcholine or Low-dose Rocuronium for Rigid Bronchoscopy: A Randomized Study
Brief Title: Muscle Relaxation for Short Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Horst Schmidt Klinik GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: HSK001; 2011_333N-MA (Registry Identifier: medical faculty of the University Mannheim)
Record Dates: First submitted 2013-07-09; First posted 2013-07-18 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2013-07

CONDITIONS: Intubating Conditions; Fasciculations; Postoperative Myalgia; Patient Satisfaction; Sore Throat
Keywords: succinylcholine; rocuronium; sugammadex; Intubating Conditions; short Procedures
MeSH Terms: conditions — Fasciculation; Patient Satisfaction; Pharyngitis | interventions — Succinylcholine; Rocuronium; Sugammadex

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Succinylcholine (Active Comparator): Patient received succinylcholine as a muscle relaxant(0.5 mg /kg)for induction of anaesthesia for rigid bronchoscopy.
  Interventions: Drug: Succinylcholine
- Rocuronium/Sugammadex (Active Comparator): Patient received rocuronium (0.25 mg/ kg) as muscle relaxant for induction of anaesthesia for rigid bronchoscopy, at the end of procedure rocuronium was reversed with sugammadex (0.5mg/kg.)
  Interventions: Drug: Rocuronium/Sugammadex
- Rocuronium (Active Comparator): Patients received rocuronium (0.25 mg /kg)as muscle relaxant for induction of anaesthesia for rigid bronchoscopy.
  Interventions: Drug: Rocuronium

INTERVENTIONS:
Drug: Succinylcholine — Anaesthesia was induced and maintained with propofol (1-2 mg/kg) and remifentanil (0.5 µg/kg). The study arm was immobilized and a dual electrode for peripheral nerve stimulation was placed over the ulnar nerve near the wrist. Neuromuscular monitoring was performed with accelerometry.The patients received succinycholine according to the study group.
  Arms: Succinylcholine
Drug: Rocuronium/Sugammadex — Anaesthesia was induced and maintained with propofol (1-2 mg/kg) and remifentanil (0.5 µg/kg). The study arm was immobilized and a dual electrode for peripheral nerve stimulation was placed over the ulnar nerve near the wrist. Neuromuscular monitoring was performed with accelerometry.The patients received rocuronium/sugammadex according to the study group.
  Arms: Rocuronium/Sugammadex
Drug: Rocuronium — Anaesthesia was induced and maintained with propofol (1-2 mg/kg) and remifentanil (0.5 µg/kg). The study arm was immobilized and a dual electrode for peripheral nerve stimulation was placed over the ulnar nerve near the wrist. Neuromuscular monitoring was performed with accelerometry.The patients received rocuronium according to the study group.
  Arms: Rocuronium

SUMMARY:
Succinylcholine is commonly used for neuromuscular relaxation for short procedures such as rigid bronchoscopy. A more modern alternative is the application of low-dose rocuronium, reversed by low-dose sugammadex. The investigators compare the intubating conditions, incidence of postoperative myalgia (POM), as well as patient satisfaction for these two muscle relaxants.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 yr
* scheduled for elective rigid bronchoscopy

Exclusion Criteria:

* known neuromuscular disease
* significant hepatic or renal dysfunction
* family history of malignant hyperthermia
* known allergy to one of the drugs used in this protocol
* pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2011-10; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Intubating condition | After induction of general anaesthesia (after 3-5 minutes)
  scoring system proposed for Good Clinical Research Practice using the following variables: conditions of inserting rigid bronchoscope, vocal cord position, and coughing

SECONDARY OUTCOMES:
Fasciculations | After application of the neuromuscular blocking agent (after 3-5 min)
  Fasciculations were graded by the investigator on the following four-point scale
  0 = no fasciculations
  1. = mild, fine fasciculations of the eyes, neck, face or fingers, without limb movement
  2. = moderate fasciculations occurring at more than two sites, or obvious limb movement
  3. = vigorous or severe, sustained and widespread fasciculations in the trunk and limbs
Postoperative Myalgia (POM) | 72 Hours after Intervention
  The severity of POM was measured using a four-point scale 0 = no myalgia
  1. = minor pain limited to one area of the body
  2. = muscle pain or stiffness noticed spontaneously by the patient, which may have required analgesic therapy
  3. = generalized, severe, or incapacitating discomfort

OTHER OUTCOMES:
Sore throat | 72 hours after intervention
  Measurement on an numeric ten point scale, the patients receive a questionaire
Patient Satisfaction | 72 Hours after intervention
  Measurement on a numeric ten point scale the patients receive a questionaire

CONTACTS AND LOCATIONS:
Overall Officials: Grietje Beck, Prof, Study Chair — Dr. Horst Schmidt Kliniken Wiesbaden Germany
Locations (1):
- Dr. Horst Schmidt Kliniken, Wiesbaden, Germany